CLINICAL TRIAL: NCT03267940
Title: A Phase 1B, Randomized, Open-Label Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) in Combination With Cisplatin Plus Gemcitabine and PEGPH20 in Combination With Atezolizumab and Cisplatin Plus Gemcitabine Compared With Cisplatin Plus Gemcitabine in Subjects With Previously Untreated, Unresectable, Locally Advanced, or Metastatic Intrahepatic and Extrahepatic Cholangiocarcinoma and Gallbladder Adenocarcinoma
Brief Title: Study of PEGPH20 With Cisplatin (CIS) and Gemcitabine (GEM); PEGPH20 With Atezolizumab (ATEZO), CIS, and GEM; and CIS and GEM Alone in Participants With Previously Untreated, Unresectable, Locally Advanced, or Metastatic Intrahepatic and Extrahepatic Cholangiocarcinoma and Gallbladder Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Halo-110-101
Record Dates: First submitted 2017-07-25; First posted 2017-08-31 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Cholangiocarcinoma Non-resectable; Cholangiocarcinoma, Intrahepatic; Cholangiocarcinoma, Extrahepatic; Gallbladder Adenocarcinoma
Keywords: Extrahepatic Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma; Gallbladder Adenocarcinoma; PEGylated Recombinant Human Hyaluronidase; PEGylated Recombinant Human Hyaluronidase with atezolizumab
MeSH Terms: conditions — Cholangiocarcinoma | interventions — PEGPH20; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Run-in Portion: PEGCISGEM (Experimental): Participants will receive 3.0 micrograms per kilogram (mcg/kg) PEGPH20 on Days 1, 8, and 15 in combination with 25 milligrams per meter square (mg/m^2) of CIS plus 1000 mg/m^2 of GEM administered on Days 2 and 9 of each 21-day cycle by intravenous (IV) infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: CIS; Drug: GEM
- Run-in Portion: PEGCISGEMATEZO (Experimental): After 6 participants from the PEGCISGEM arm are treated for at least 1 cycle without significant toxicities, new participants will be enrolled in this arm to receive 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: CIS; Drug: GEM; Drug: Atezolizumab
- Expansion Portion: PEGCISGEM (Experimental): After the Investigators and the Sponsor considers the study treatment with PEGCISGEM during the Run-in portion safe and tolerable, new participants will be enrolled to receive 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 25 mg/m^2 CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: CIS; Drug: GEM
- Expansion Portion: PEGCISGEMATEZO Twice Weekly (Experimental): After the Investigators and the Sponsor considers the study treatment with PEGCISGEM during the Run-in portion safe and tolerable, new participants will be enrolled to receive 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: CIS; Drug: GEM; Drug: Atezolizumab
- Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly (Experimental): After the implementation of Protocol Amendment #3 and as communicated to the Investigators via a letter dated 22 March 2019, participants will receive 3.0 mcg/kg PEGPH20 on Days 1, 4, 8, 11, 15 and 18 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 Cycle 1) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of Cycle 1 (cycle length = 21 days) by IV infusion. Participants will receive 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle from Cycle 2 and beyond by IV infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: PEGPH20; Drug: CIS; Drug: GEM; Drug: Atezolizumab
- Expansion Portion: CISGEM (Active Comparator): After the Investigators and the Sponsor considers the study treatment with PEGCISGEM during the run-in portion safe and tolerable, new participants will be enrolled to receive 25 mg/m^2 CIS and 1000 mg/m^2 GEM on Days 1 and 8 of each 21-day cycle by IV infusion. Treatment will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.
  Interventions: Drug: CIS; Drug: GEM

INTERVENTIONS:
Drug: PEGPH20 — PEGPH20 will be administered as per the schedule specified in the respective arms.
  Arms: Expansion Portion: PEGCISGEM; Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly; Expansion Portion: PEGCISGEMATEZO Twice Weekly; Run-in Portion: PEGCISGEM; Run-in Portion: PEGCISGEMATEZO
Drug: CIS — CIS will be administered as per the schedule specified in the respective arms.
Drug: GEM — GEM will be administered as per the schedule specified in the respective arms.
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in the respective arms.
  Arms: Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly; Expansion Portion: PEGCISGEMATEZO Twice Weekly; Run-in Portion: PEGCISGEMATEZO

SUMMARY:
The study is being conducted to assess the safety and tolerability of (1) PEGPH20 in combination with CIS and GEM (PEGCISGEM), and (2) PEGPH20 in combination with CIS, GEM, and atezolizumab (PEGCISGEMATEZO) compared with (3) cisplatin and gemcitabine (CISGEM).

DETAILED DESCRIPTION:
The study will have a Run-in portion and an Expansion portion. The Run-in portion will be used to evaluate the safety profile of the PEGCISGEM and PEGCISGEMATEZO treatments prior to evaluating the efficacy and safety of PEGCISGEM and PEGCISGEMATEZO treatments compared with CISGEM treatment in the Expansion portion of the study. Treatment in both portions of the study will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

For both portions of the study, participants must satisfy all of the following inclusion criteria to be enrolled in the study:

* Written Institutional Review Board/Ethics Committee-approved informed consent form (ICF), signed by participant or legally authorized representative.
* Participants must be determined to have histologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of the intra- and/or extra-hepatic bile ducts and/or gallbladder. Participants must have sufficient tissue with architectural integrity, including tumor and associated stroma, available for retrospective biomarker testing.
* One or more lesions measurable on computed tomography (CT) scan/magnetic resonance imaging (MRI) scan per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1).
* Participants having Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Life expectancy ≥3 months.
* Males and females aged ≥18 years.
* Screening clinical laboratory values within pre-determined parameters
* Female participants of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days before Day 1 (first dose of study medication).
* For WOCBP and for men, agreement to use a highly effective contraceptive method from the time of screening throughout the study until 5 months (WOCBP) or 6 months (men) after administration of the last dose of any study medication. Highly effective contraceptive methods consist of prior sterilization, intrauterine device (IUD), intrauterine hormone releasing system (IUS), oral or injectable contraceptives, barrier methods, and/or true sexual abstinence.

Exclusion Criteria:

Participants are ineligible for enrollment if they meet any of the following exclusion criteria:

* Clinical evidence of deep vein thrombosis or pulmonary embolism present during the screening period
* New York Heart Association Class III or IV cardiac disease, atrial fibrillation, unstable angina, or myocardial infarction within the past 12 months before screening.
* Participants with known brain metastases
* History of cerebrovascular accident or transient ischemic attack
* History of active bleeding within the last 3 months prior to screening requiring transfusion.
* Participants must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for treatment of metastatic or locally advanced disease.
* Intolerance to non-steroidal anti-inflammatory drugs (NSAIDs).
* Active hepatitis B virus (HBV) infection, defined as having a positive hepatitis B surface antigen (HBsAg) test at screening
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test at screening
* History of:

  1. Idiopathic pulmonary fibrosis, organizing pneumonia (for example, bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
  2. Or known cases of hepatobiliary diseases (for example, primary biliary cholangitis, primary sclerosing cholangitis, history of immune-mediated cholangitis);

     Participants with cholangitis attributed to infectious etiology (for example, ascending cholangitis, bacterial cholangitis) are eligible if the infection has been fully resolved prior to the screening visit.
  3. Or known cases of drug-induced hepatobiliary toxicities.
* Active or history of autoimmune diseases
* Uncontrolled hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Medical, Regulatory and Drug Safety, Study Director — Halozyme Therapeutics
Locations (36):
- United States (26):
  - Mayo Clinic of Arizona, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - City of Hope, Duarte, California
  - Scripps, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Division of Hematology-Oncology, Department of Medicine UC Irvine Health, Orange, California
  - UC Davis, Sacramento, California
  - UCLA - David Geffen School of Medicine, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Yale Cancer Center, New Haven, Connecticut
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - UT Health Cancer Center, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert Hospital And Medical College, Milwaukee, Wisconsin
- South Korea (7):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-Gu
  - Asan Medical Center, Seoul, Songpa-gu
- Thailand (3):
  - Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Muang
  - King Chulalongkorn Memorial Hospital, Bangkok, Patumwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 portions: Run-in portion and Expansion portion.
Pre-assignment Details: The study was terminated prematurely by the Sponsor due to stopping the clinical development of PEGPH20 in all indications based on negative pivotal data in metastatic pancreatic cancer.
Groups:
- Run-in Portion: PEGCISGEM: Participants received 3.0 micrograms per kilogram (mcg/kg) PEGPH20 on Days 1, 8, and 15 in combination with 25 milligrams per meter square (mg/m^2) of cisplatin (CIS) plus 1000 mg/m^2 of gemcitabine (GEM) administered on Days 2 and 9 of each 21-day cycle by intravenous (IV) infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity. (Maximum exposure: 190 days)
- Run-in Portion: PEGCISGEMATEZO: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg atezolizumab (ATEZO) (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity. (Maximum exposure: 508 days)
- Expansion Portion: PEGCISGEM: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 25 mg/m^2 CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (Maximum exposure: 421 days).
- Expansion Portion: PEGCISGEMATEZO Twice Weekly: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (Maximum exposure: 416 days).
- Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 4, 8, 11, 15 and 18 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 Cycle 1) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of Cycle 1 (cycle length = 21 days) by IV infusion. Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle from Cycle 2 and beyond by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (Maximum exposure: 59 days).
- Expansion Portion: CISGEM: Participants received 25 mg/m^2 CIS and 1000 mg/m^2 GEM on Days 1 and 8 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (Maximum exposure: 218 days).
Period: Run-in Portion (Max. Exposure: 508 Days)
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Started | 9 | 9 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 9 | 9 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 0 | 0 | 0 | 0
Not Completed | 8 | 7 | 0 | 0 | 0 | 0
Not completed — Investigator or Sponsor Decision | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Terminated Study | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 7 | 3 | 0 | 0 | 0 | 0
Period: Expansion (Maximum Exposure: 421 Days)
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Started | 0 | 0 | 24 | 22 | 11 | 10
Received at Least 1 Dose of Study Drug | 0 | 0 | 24 | 22 | 11 | 10
Completed | 0 | 0 | 3 | 0 | 1 | 0
Not Completed | 0 | 0 | 21 | 22 | 10 | 10
Not completed — Other than specified | 0 | 0 | 0 | 3 | 2 | 0
Not completed — Investigator or Sponsor Decision | 0 | 0 | 2 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 1 | 1
Not completed — Sponsor Terminated Study | 0 | 0 | 7 | 4 | 5 | 3
Not completed — Death | 0 | 0 | 10 | 13 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled population included all participants enrolled in the Run-in portion and the Expansion portion of the study.
Groups:
- Run-in Portion: PEGCISGEM: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 25 mg/m^2 of CIS plus 1000 mg/m^2 of GEM administered on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity. (Maximum exposure: 190 days)
- Run-in Portion: PEGCISGEMATEZO: Participants received 3.0 mcg/kg PEGPH20 on Days 1, 8, and 15 in combination with 1200 mg ATEZO (administered 1 to 3 hours after PEGPH20 on Day 1 of each 21-day cycle) plus 25 mg/m^2 of CIS and 1000 mg/m^2 GEM on Days 2 and 9 of each 21-day cycle by IV infusion. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity. (Maximum exposure: 508 days)
- Total: Total of all reporting groups
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM | Total
Number analyzed (Participants) | 9 | 9 | 24 | 22 | 11 | 10 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 15 | 10 | 4 | 6 | 45
  >=65 years | 2 | 6 | 9 | 12 | 7 | 4 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 13 | 8 | 6 | 8 | 43
  Male | 3 | 7 | 11 | 14 | 5 | 2 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 9 | 8 | 24 | 21 | 11 | 8 | 81
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 9 | 7 | 3 | 4 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 5 | 4 | 14 | 14 | 7 | 6 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Run-in Portion: Number of Participants With Adverse Events (AEs)
Description: An AE is any unfavorable or unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product (for example, study drug), whether or not considered related to the pharmaceutical product. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through 30 days after the end of treatment visit (maximum exposure: 508 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

2. Primary Outcome: Run-in Portion: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters (Hematology and Blood Chemistry)
Description: Laboratory parameters evaluation included hematology (hemoglobin, hematocrit, red blood cell count, white blood cell [WBC] count, neutrophils [ANC], lymphocytes, monocytes, eosinophils, basophils, granulocytes, mean corpuscular hemoglobin, mean corpuscular volume, and platelet count) and blood chemistry (glucose, blood urea nitrogen [BUN], albumin, total bilirubin, alkaline phosphatase, aspartate aminotransferase [AST], alanine aminotransferase [ALT], electrolytes [including sodium, potassium, calcium, magnesium, chloride, and bicarbonate], and creatinine) evaluation. Clinical significance was defined as per Investigator's discretion. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 508 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

3. Primary Outcome: Run-in Portion: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) and Vital Signs
Description: Clinical significance of ECGs was defined as per Investigator's discretion. Assessment of vital signs was to include the measurement of blood pressure (systolic and diastolic), pulse, respiratory rate, and body temperature. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 508 days)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Run-in Portion: Number of Participants With AEs Leading to Dose Reduction or Interruption of Any Study Medication
Description: Number of participants with AEs leading to dose reduction or interruption of any study medication (PEGPH20, CIS, GEM, or ATEZO) was reported. An AE is any unfavorable or unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product (for example, study drug), whether or not considered related to the pharmaceutical product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 508 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO
Number analyzed (Participants) | 9 | 9
Participants | 6 | 7

5. Primary Outcome: Expansion Portion: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1: Percentage of Participants With Objective Response
Description: ORR was defined as percentage of participants who achieved either a complete response (CR) or partial response (PR). CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the date of first documented progression of disease or date of death from any cause, whichever came first (maximum exposure: 421 days)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Run-in Portion: ORR Based on RECIST v1.1: Percentage of Participants With Objective Response
Description: ORR was defined as percentage of participants who achieved either a CR or PR. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the date of first documented progression of disease or date of death from any cause, whichever came first (maximum exposure: 508 days)
Population: Data for this outcome measure was not Collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Expansion Portion: Duration of Response (DOR) Based on RECIST v1.1
Description: DOR was considered the time from date of the first CR or PR until the date of first documentation of disease progression or date of death based on RECIST v1.1 for target lesions assessed by MRI/CT scans, as determined by independent radiologic review. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: From date of the first CR or PR until the date of first documentation of disease progression or date of death, whichever came first (maximum exposure: 421 days)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Expansion Portion: Progression-Free Survival (PFS) Based on RECIST v1.1
Description: PFS was based on RECIST v1.1 for target lesions assessed by MRI/CT scans, as determined by independent radiologic review and was defined as the time from randomization to radiological disease progression or death. Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on or prior to the current assessment (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of greater than or equal to (≥) 5 mm.
Time Frame: From date of randomization until date of progressive disease or death from any cause, whichever came first (maximum exposure: 421 days)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Expansion Portion: Disease Control Rate (DCR) Based on RECIST v1.1: Percentage of Participants With CR, PR or Stable Disease (SD)
Description: DCR was defined as the percentage of participants with CR, PR, or SD based on RECIST v1.1 for target lesions assessed by MRI/CT scans, as determined by independent radiologic review. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
Time Frame: as for outcome 8
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Expansion Portion: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: From randomization until death from any cause (maximum exposure: 421 days)
Population: This data was not collected as an endpoint but all deaths due to any cause are reported in the AE module.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Expansion Portion: OS by PD-L1 Expression Levels
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: From randomization until death from any cause (maximum exposure: 421 days)
Population: This data was not collected as an endpoint but all deaths due to any cause are reported in the AE module.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Expansion Portion: Number of Participants With AEs
Description: An AE is any unfavorable or unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product (for example, study drug), whether or not considered related to the pharmaceutical product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 421 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 24 | 22 | 11 | 10
Participants | 24 | 22 | 10 | 10

13. Secondary Outcome: Expansion Portion: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters (Hematology and Blood Chemistry)
Description: Laboratory parameters evaluation included hematology (hemoglobin, hematocrit, red blood cell count, WBC count, neutrophils [ANC], lymphocytes, monocytes, eosinophils, basophils, granulocytes, mean corpuscular hemoglobin, mean corpuscular volume, and platelet count) and blood chemistry (glucose, BUN, albumin, total bilirubin, alkaline phosphatase, AST, ALT, electrolytes [including sodium, potassium, calcium, magnesium, chloride, and bicarbonate], and creatinine) evaluation. Clinical significance was defined as per Investigator's discretion. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 421 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 24 | 22 | 11 | 10
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Expansion Portion: Number of Participants With Clinically Significant Abnormalities in ECG and Vital Signs
Description: as for outcome 3
Time Frame: From first exposure to study drug through the end of treatment visit (maximum exposure: 421 days)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Expansion Period: Number of Participants With AEs Leading to Dose Reduction or Interruption of Any Study Medication
Description: as for outcome 4
Time Frame: From first exposure to study drug through 30 days after the end of treatment visit (maximum exposure: 421 days)
Population: Safety population included all participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 24 | 22 | 11 | 10
Participants | 16 | 21 | 4 | 7

16. Secondary Outcome: Run-in and Expansion Portion : Maximum Observed Plasma Concentration (Cmax) of PEGPH20, ATEZO, GEM, and CIS
Description: Plasma pharmacokinetic (PK) data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: PEGPH20 and ATEZO: Cycle 1: multiple timepoints on Days 1, 2, 8, 9, 15; ATEZO: Day 1 of subsequent cycles and end of treatment (EOT) (maximum exposure: 508 days for run-in and 421 days for expansion); CIS and GEM: Cycle 1: multiple timepoints on Days 2,9
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Run-in and Expansion Portion : Minimum Observed Plasma Concentration (Cmin) of PEGPH20 and ATEZO
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: PEGPH20 and ATEZO: Treatment Cycle 1: multiple timepoints on Days 1, 2, 8, 9, and 15; ATEZO: Day 1 of subsequent cycles and EOT visit (7 days after last 21-day cycle) (maximum exposure: 508 days for run-in portion and 421 days for expansion portion)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Run-in and Expansion Portion : Elimination Rate Constant (Kel) of PEGPH20
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: Cycle 1: multiple timepoints on Days 1, 2, 8, 9, and 15
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Run-in and Expansion Portion : Terminal Elimination Plasma Half-life (t1/2) of PEGPH20, ATEZO, GEM, and CIS
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: PEGPH20 and ATEZO: Cycle 1: multiple timepoints on Days 1, 2, 8, 9, 15; ATEZO: Day 1 of subsequent cycles and EOT visit (maximum exposure: 508 days for run-in and 421 days for expansion portion); CIS and GEM: Cycle 1: multiple timepoints on Days 2, 9
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Run-in and Expansion Portion : Clearance (CL) of PEGPH20, ATEZO, GEM, and CIS
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: as for outcome 19
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Run-in and Expansion Portion : Volume of Distribution (Vd) of PEGPH20, ATEZO, GEM, and CIS
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: as for outcome 19
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Run-in and Expansion Portion: Area Under the Concentration Time Curve (AUC) of PEGPH20, ATEZO, GEM, and CIS
Description: PK data were planned to be analyzed using a noncompartmental analysis approach.
Time Frame: as for outcome 19
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first exposure to study drug through 30 days after end of treatment visit (maximum exposure: 508 days for run-in portion and 421 days for expansion portion)
Description: Safety population included all participants who received any study medication.
Arm/Group | Run-in Portion: PEGCISGEM | Run-in Portion: PEGCISGEMATEZO | Expansion Portion: PEGCISGEM | Expansion Portion: PEGCISGEMATEZO Twice Weekly | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly | Expansion Portion: CISGEM
All-Cause Mortality (participants affected / at risk) | 7/9 | 3/9 | 10/24 | 13/22 | 0/11 | 6/10
Serious Adverse Events (participants affected / at risk) | 6/9 | 2/9 | 11/24 | 16/22 | 7/11 | 4/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 24/24 | 22/22 | 10/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Run-in Portion: PEGCISGEM (N=9) | Run-in Portion: PEGCISGEMATEZO (N=9) | Expansion Portion: PEGCISGEM (N=24) | Expansion Portion: PEGCISGEMATEZO Twice Weekly (N=22) | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly (N=11) | Expansion Portion: CISGEM (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 5 | 2 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 4 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Systemic immune activation (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis infective (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ovarian necrosis (Reproductive system and breast disorders) | 0/6 | 0/2 | 1/13 | 0/8 | 0/6 | 0/8 — This is a sex-specific adverse event that only affects female participants.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Run-in Portion: PEGCISGEM (N=9) | Run-in Portion: PEGCISGEMATEZO (N=9) | Expansion Portion: PEGCISGEM (N=24) | Expansion Portion: PEGCISGEMATEZO Twice Weekly (N=22) | Expansion Portion: PEGCISGEMATEZO Once Weekly/Twice Weekly (N=11) | Expansion Portion: CISGEM (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 12 | 15 | 3 | 8
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 3 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 5 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 5 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 10 | 5 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 4 | 10 | 8 | 3 | 5
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 9 | 9 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 18 | 11 | 3 | 9
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3 | 12 | 7 | 1 | 5
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 1 | 2 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 4 | 0 | 1
Fatigue (General disorders) | 5 | 8 | 15 | 13 | 2 | 6
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 5 | 10 | 10 | 3 | 3
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 6 | 11 | 3 | 5
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 4 | 6 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 6 | 8 | 3 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 3 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 4 | 2 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 3 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Granulocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Grip strength decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 4 | 7 | 8 | 2 | 2
Platelet count decreased (Investigations) | 1 | 3 | 5 | 8 | 2 | 5
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 4 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 5 | 9 | 2 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 6 | 5 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 9 | 7 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 5 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 11 | 8 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 8 | 7 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 3 | 5 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 3 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2 | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 5 | 1 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 4 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 5 | 7 | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/6 | 0/2 | 1/13 | 0/8 | 0/6 | 0/8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 4 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 3 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prurit (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 3 | 2 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the Sponsor due to stopping the clinical development of PEGPH20 in all indications based on negative pivotal data in metastatic pancreatic cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03267940/Prot_000.pdf